CLINICAL TRIAL: NCT02612584
Title: Clinical Efficacy of the Pinhole Soft Contact Lenses for Correcting Presbyopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1-2015-0015
Record Dates: First submitted 2015-11-18; First posted 2015-11-24 (Estimated); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pinhole soft contact lens (Experimental)
  Interventions: Device: Pinhole Soft Contact Lens apply for presbyopia

INTERVENTIONS:
Device: Pinhole Soft Contact Lens apply for presbyopia

SUMMARY:
For correct of presbyopia, in this study, the investigators have recruited subjects who aged 45~65 years with presbyopia and do not have any other ocular disease(ex, ocular surface disease, corneal dystrophy, retinal disorders, etc.). All participants will underwent ophthalmic examination including manifest refraction, uncorrected distance visual acuity (UDVA), uncorrected near visual acuity (UNVA), corrected distance visual acuity (CDVA), corrected near visual acuity(CNVA), Goldmann visual field test, depth of focus Contrast sensitivity test, slit-lamp examination, topography with scheimp flug device(OCULUS pentacam ®) OSDI(ocular surface disease index) and Questionnaire about visual function and ocular symptoms. Apply pinhole soft contact lens (eyelike NoanPinhole ® , seoul, south Korea, Koryo Eyetech) on non-dominant eye of participants and/or soft contact lens for distance vision on dominant eye of participants. The investigators recommend use of pinhole contact lens at least 3 hours in a day for 1 week. And, participant will underwent the all ophthalmic examination same above 2 weeks after first apply of pinhole contact lens. The investigators will compare ophthalmic parameters mentioned above before and after wearing pinhole contact lens and evaluate the efficacy and safety of pinhole soft contact lens for correcting presbyopia.

ELIGIBILITY:
Inclusion Criteria:

* Age, 45~65 years with presbyopia

Exclusion Criteria:

* Patients with anterior segment pathology,
* Patients with previous intraocular or corneal surgery,
* Patients with severe cataracts,
* Patients with corneal abnormalities( including endothelial dystrophy, recurrent corneal erosion, etc.),
* Patients with history of chronic dry eye, macular degeneration,
* Patients with retinal detachment, or any other fundus pathology

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-01-01; Primary Completion 2016-11-15 (Actual); Study Completion 2016-11-15 (Actual)

PRIMARY OUTCOMES:
Corrected (with pinhole contact lens) Near Vision Acuity | 2 weeks after first apply of pinhole contact lens
Defocusing curve | 2 weeks after first apply of pinhole contact lens

SECONDARY OUTCOMES:
Corneal erosion grade(oxford score) | 2 weeks after first apply of pinhole contact lens
OSDI(ocular surface disease index) | 2 weeks after first apply of pinhole contact lens
Visual field test | 2 weeks after first apply of pinhole contact lens
Contrast sensitivity test | 2 weeks after first apply of pinhole contact lens

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, Yonsei Univeristy College of Medicine, Seoul, South Korea

REFERENCES:
- [Background] Schwiegerling J. Predicting clinical visual acuity of presbyopia treatments. J Refract Surg. 2010 Jan;26(1):66-70. doi: 10.3928/1081597X-20101215-11. PMID 20199016
- [Background] Garcia-Lazaro S, Ferrer-Blasco T, Radhakrishnan H, Albarran-Diego C, Montes-Mico R. Visual comparison of an artificial pupil contact lens to monovision. Optom Vis Sci. 2012 Jul;89(7):E1022-9. doi: 10.1097/OPX.0b013e31825da324. PMID 22729169
- [Background] Charman WN. Developments in the correction of presbyopia I: spectacle and contact lenses. Ophthalmic Physiol Opt. 2014 Jan;34(1):8-29. doi: 10.1111/opo.12091. Epub 2013 Nov 10. PMID 24205890
- [Background] Callina T, Reynolds TP. Traditional methods for the treatment of presbyopia: spectacles, contact lenses, bifocal contact lenses. Ophthalmol Clin North Am. 2006 Mar;19(1):25-33, v. doi: 10.1016/j.ohc.2005.09.006. PMID 16500526